CLINICAL TRIAL: NCT03346863
Title: Predictors for Recurrence of Atrial Fibrillation After Electrical Cardioversion
Acronym: PRE-ELECTRIC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Vestre Viken Hospital Trust (Other)
Collaborators: Oslo University Hospital (Other); Lund University (Other)
Responsible Party: Sponsor
Other Study IDs: PRE-ELECTRIC 2017/1604
Record Dates: First submitted 2017-11-14; First posted 2017-11-17 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Atrial Fibrillation
Keywords: Electrical Cardioversion
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, EDTA Plasma, Citrated Plasma, EDTA Whole Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In patients with persistent atrial fibrillation (AF), electrical cardioversion is very effective in restoring sinus rhythm if modern, biphasic cardioverters are used. However, approximately 50 per cent of the successfully cardioverted patients experience a recurrence of AF within a few weeks. Therefore, valid predictors for AF recurrence would be of great clinical relevance, to avoid unnecessary procedures.

In the PRE-ELECTRIC study, we will investigate the predictive value of potential new biomarkers with respect to AF recurrence within 30 days after electrical cardioversion. We will investigate serum and plasma biomarkers, electrocardiological markers and echocardiographic variables in this respect. The study will be undertaken as a prospective cohort study at Bærum Hospital, Vestre Viken Hospital Trust, with national and international collaborators.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years referred for electrical cardioversion for persistent atrial fibrillation
* Signed, informed consent

Exclusion Criteria:

* Patients < 18 years
* Patients with paroxysmal atrial fibrillation
* Patients unwilling to participate or without consent competence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients > 18 years referred for electrical cardioversion for ECG-documented persistent atrial fibrillation.
Sampling Method: Non-Probability Sample
Enrollment: 270 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Atrial fibrillation recurrence | 30 days after electrical cardioversion
  ECG-documented atrial fibrillation recurrence after successful cardioversion

CONTACTS AND LOCATIONS:
Locations (1):
- Bærum Hospital, Vestre Viken, Sandvika, Bærum, Norway

IPD SHARING:
Plan to Share IPD: No